CLINICAL TRIAL: NCT02563639
Title: APAF Apixaban in Atrial Fibrillation Registry
Brief Title: Apixaban in Atrial Fibrillation Registry
Acronym: APAF
Status: Completed | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-404
Record Dates: First submitted 2015-09-21; First posted 2015-09-30 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
Keywords: newly diagnosed; paroxysmal; persistent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective of the registry is to assess the use of antithrombotic therapies and adherence to guidelines in patients with non-valvular atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) confers a substantial risk of mortality and morbidity from stroke and thromboembolism, and this common cardiac arrhythmia represents a major healthcare burden in Europe. Stroke prevention is central to the management of AF patients, with oral anticoagulation (OAC) using well-controlled adjusted dose vitamin K antagonists or novel OACs being recommended for patients with AF with ≥1 stroke risk factors. Also, the 2012 focused update of the ESC guidelines strongly advocates a clinical practice shift so that the initial decision step now is the identification of 'truly low risk' patients, essentially those age<65 without any stroke risk factors (both male and female), who do not need any antithrombotic therapy. The ESC guidelines only recommend use of the CHA2DS2-VASc score for stroke risk assessment, and the 'low risk' patients are defined as those with a CHA2DS2-VASc score=0 (males) or score=1 (females). Subsequent to this initial step of identifying the low risk patients, effective stroke prevention (which is essentially OAC) can then be offered to AF patients with ≥1 stroke risk factors, with treatment decisions made in consultation with patients and incorporating their preferences. Despite these recommendations, a substantial number of patients with AF is not treated with OAC. On the other hand, patients with AF and low risk are being "overtreated", receiving OAC despite a CHADS-VASc score of 0. Therefore, this registry will determine, if patients with non-valvular AF are treated ac-cording to current guidelines.

Apixaban is an oral factor Xa inhibitor, which has been tested in a number of indications. In the AVERROES study in patients with non-valvular atrial fibrillation deemed not suitable for treatment with a vitamin-K antagonist apixaban compared to aspirin reduced the incidence of stroke and systemic embolism without increasing bleeding complications. In the large ARISTOTELE study apixaban was superior to warfarin, it re-duced the primary endpoint of stroke and systemic embolism caused less bleeding and reduced all-cause mortality. Subsequently apixaban has been approved by the European health authorities for the use in patients with atrial fibrillation. It is therefore of interest to determine use of apixaban in real life with respect to patient selection, adherence to therapy and midterm efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Non-valvular atrial fibrillation
* In hospitals or specialized or non-specialised office-based centres
* Written informed consent for participation in observational study (incl. telephone follow-ups)
* Not simultaneously participating in any randomized trial

Exclusion Criteria: No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation (newly diagnosed, paroxysmal, permanent or persistent)
Sampling Method: Non-Probability Sample
Enrollment: 5015 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Comparison of antithrombotic therapy for atrial fibrillation: Prescribed drugs | 12 months
  Name of antithrombotic drug

SECONDARY OUTCOMES:
Safety of Apixaban as assessed by MACCE, Haemorrhagic complications, Ischemic clinical events, Stroke, Systemic embolism, Hospitalisations for stroke, cardiac reasons or bleeding complications | 12 months
  * MACCE (death / MI / stroke)
  * Haemorrhagic complications (major / minor bleeding)
  * Ischemic clinical events (non-fatal MI, cardiac death, etc.)
  * Stroke (ischemic, haemorrhagic)
  * Systemic embolism
  * Hospitalisations for stroke, cardiac reasons or bleeding complications
Subjective Quality of Life | 12 months
  Questionnaire (EQ-5D-5L)
Comparison of antithrombotic therapy for atrial fibrillation: Dose of drugs | 12 months
  Dose of antithrombotic drug
Comparison of antithrombotic therapy for atrial fibrillation: Duration of treatment | 12 months
  Duration of treatment [months]
Comparison of antithrombotic therapy for atrial fibrillation: Contraindications for anticoagulation | 12 months
  Relative and absolute contraindications to anticoagulation at baseline and history
Comparison of antithrombotic therapy for atrial fibrillation:Selection of anticoagulant | 12 months
  Basis for the selection of the anticoagulant

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Zeymer, Prof. Dr., Principal Investigator — Klinikum Ludwigshafen
Locations (1):
- Klinikum Ludwigshafen, Ludwigshafen, Germany